CLINICAL TRIAL: NCT00505895
Title: A Randomized Phase II Trial of Fludarabine/Melphalan 140 VS. Fludarabine/Melphalan 100 Followed By Allogeneic Peripheral Blood Stem Cell or Bone Marrow Transplantation for Patients With Multiple Myeloma
Brief Title: FM 140 vs FM100 Study in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID01-518
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Fludarabine; Fludara; Fludarabine Phosphate; Melphalan; Alkeran; Stem Cell Infusion; Stem Cell Transfusion; SCT; Allogeneic Peripheral Blood Stem Cell Transfusion; APBSCT; Bone Marrow Transplantation; BMT; Rituxan; Rituximab; FM140; FM100
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; fludarabine; fludarabine phosphate; Bone Marrow Transplantation; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine + Melphalan + Stem Cell Infusion (Experimental): Fludarabine 30 mg/m^2 intravenous (IV) daily over 30 minutes for 4 Days (Beginning Day -4).
  Melphalan 140 mg/m^2 IV over 20 minutes on Day -1. Stem Cell Infusion on Day 0. Rituximab 375 mg/m^2 IV infused starting on day -5.
  Interventions: Drug: Melphalan; Drug: Fludarabine; Procedure: Stem Cell Infusion; Drug: Rituximab
- Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion (Experimental): Fludarabine 30 mg/m^2 intravenous daily over 30 minutes for 4 Days (Beginning Day -4).
  Lower-Dose Melphalan 100 mg/m^2 intravenous over 20 minutes on Day -1. Stem Cell Infusion on Day 0. Rituximab 375 mg/m^2 intravenous infused starting on day -5.
  Interventions: Drug: Melphalan; Drug: Fludarabine; Procedure: Stem Cell Infusion; Drug: Rituximab

INTERVENTIONS:
Drug: Melphalan — Arm 1 = 140 mg/m^2 intravenous over 20 Minutes on Day -1; Arm 2 = 100 mg/m^2 intravenous over 20 Minutes on Day -1.
  Other Names: Alkeran
Drug: Fludarabine — 30 mg/m^2 intravenous daily over 30 Minutes for 4 Days (Beginning Day -4).
  Other Names: Fludara; Fludarabine Phosphate
Procedure: Stem Cell Infusion — Stem Cell Infusion on Day 0.
  Other Names: Allogeneic Peripheral Blood Stem Cell Transfusion; APBSCT; Bone Marrow Transplantation; BMT
Drug: Rituximab — 375 mg/m^2 intravenous on Day -5, +2 +9 and +16.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if there is a difference in transplant outcomes between two different doses of melphalan given in combination with fludarabine followed by transfusion of a related or unrelated volunteer donor's peripheral blood or bone marrow progenitor cells (allogeneic stem cell transplant) in patients with multiple myeloma. This study will also look at whether treatment with a antibody called rituximab against a specific type of lymphocyte (B cell) will reduce the risks of developing graft versus host disease after transplant. The safety of these treatments will also be compared.

DETAILED DESCRIPTION:
Fludarabine is a chemotherapy drug that is used in various diseases. Melphalan is a chemotherapy drug that has been widely used in the treatment of multiple myeloma for many years.

Before beginning therapy, patients will have a complete work-up. This includes a bone marrow aspiration and biopsy, bone survey, blood tests, and tests to check the heart and lung function. All patients will receive tacrolimus and methotrexate to prevent graft-versus-host disease.

Patients in this study will be randomly picked (as in the toss of a coin) to be in one of two treatment groups. There is an equal chance that a patient will be in either group.

Patients in the first group will receive fludarabine through the vein every day for four days. On the fourth day, patients will receive a dose of melphalan through the vein over 20 minutes. On the following day, patients will receive the donor cells as an infusion through their catheter.

Patients in the second group will receive fludarabine through the vein every day for four days. Patients in this group will receive a lower dose of melphalan through the vein over 20 minutes. After the last dose of fludarabine, patients will receive the donor cells as an infusion through their catheter the next day.

If you have an unrelated or a mismatched donor, you will receive the drug ATG (Thymoglobulin) by vein over 6 hours on Days -3, -2, and -1 (the 3 days before the transplant), to prevent graft versus host disease (GVHD) and to help engraftment.

Patients in both group will be receiving the monoclonal antibody called rituximab weekly starting on the fifth day before the stem cell transplant for a total of 4 doses.

Patients will remain in the hospital for about 4-6 weeks and in Houston Medical Center area at least 100 days after transplantation.

Patients whose disease gets worse will be taken off study. These patients will continue to be followed for survival.

This is an investigational study. All of the drugs used in this study are commercially available. The FDA has approved melphalan for the treatment of myeloma. Fludarabine is not approved for the treatment of myeloma but has been used for years as a way to prepare patients for transplant. About 30 to 60 patients will take part in this study. About 45 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Multiple Myeloma in any of the following disease categories: a) Primary Refractory considered poor candidate for autologous transplant, b) Remission Consolidation in patients with Chromosome 13 abnormalities or plasma cell leukemia, c) All relapsing patients.
2. Age up to 70 years.
3. Related or unrelated donor who is HLA-compatible in at least 9/10 alleles (A,B, C, DRB1 and DQ) by molecular techniques.
4. Zubrod Performance Score (PS)<2.
5. Life expectancy is not severely limited by concomitant illness. Left ventricular ejection fraction >40%. No uncontrolled arrhythmias or symptomatic cardiac disease. Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lungs for carbon monoxide (DLCO) >40%.
6. Patient and donor or guardian willing and able to sign informed consent.

Exclusion Criteria:

1) Patients with active central nervous system (CNS) disease are ineligible for this study as documented by clinical symptoms and/or testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 18, 2002 to July 27, 2011. All recruitment done in a medical clinical setting.
Pre-assignment Details: Of the 52 participants enrolled, two were not included due to one patient experiencing pulmonary complication and another not completing the study follow up requirement.
Groups:
- Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion: Fludarabine 30 mg/m^2 IV daily over 30 minutes for 4 Days (Beginning Day -4).
  Lower-Dose Melphalan 100 mg/m^2 IV over 20 minutes on Day -1. Stem Cell Infusion on Day 0. Rituximab 375 mg/m^2 IV infused starting on day -5.
Period: Overall Study
Arm/Group | Fludarabine + Melphalan + Stem Cell Infusion | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fludarabine + Melphalan + Stem Cell Infusion | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Median (Full Range); unit: years] | 52 [32 to 64] | 53 [36 to 64] | 53 [32 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 19 | 11 | 30
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Engraftment at Day 100
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Fludarabine + Melphalan + Stem Cell Infusion | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion
Number analyzed (Participants) | 27 | 23
participants | 27 | 23

2. Secondary Outcome: Acute Grade II-IV Graft Versus Host Disease (GVHD)
Description: Effects of Rituximab as measured by percentage of participants with Acute and Chronic Graft Versus Host Disease (GVHD) incidences after allogeneic transplantation. GVHD occurring anytime after day 90 post transplant was considered chronic GVHD; otherwise it was considered acute GVHD. Acute GVHD status defined as GVHD with maximum grade ≥2. Clinical grading of Acute GVHD (Thomas et al., New England Journal of Medicine (NEJM), 229:895, 1975): Grade 1 to 4.
Time Frame: GVHD grading weekly during first 100 days; Annual examinations for nine year study period
Population: For the acute GVHD analysis, only 48 patients' data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Fludarabine + Melphalan + Stem Cell Infusion | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion
Number analyzed (Participants) | 27 | 23
percentage of participants
  Acute GVHD | 22 | 21
  Chronic GVHD | 29 | 48

ADVERSE EVENTS:
Time Frame: The end of active treatment was the day of the drug administration of Rituximab on Day+16. Study participation was from baseline to 100 days after transplantation. Overall study period was March 2002 to May 2013.
Arm/Group | Fludarabine + Melphalan + Stem Cell Infusion | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion
Serious Adverse Events (participants affected / at risk) | 23/27 | 16/23
Other Adverse Events (participants affected / at risk) | 8/27 | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Melphalan + Stem Cell Infusion (N=27) | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion (N=23)
Death (General disorders) | 23 (23) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection (Investigations) | 3 (5) | 6 (14)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Total Bilirubin Level Change (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Secondary graft failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 0 (0) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Melphalan + Stem Cell Infusion (N=27) | Fludarabine + Lower-Dose Melphalan + Stem Cell Infusion (N=23)
Fever (Infections and infestations) | 3 (3) | 3 (3)
Volume overload (General disorders) | 1 (1) | 3 (3)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (8) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 2 (3)
Dysarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 0 (0) | 2 (2)
Elevated ALT (Hepatobiliary disorders) | 0 (0) | 2 (2)
Lethargy (General disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No